CLINICAL TRIAL: NCT07100197
Title: EEG-TMS Intervening Against Postoperative Delirium in Elderly Patients: A Randomized Clinical Trial
Brief Title: EEG-TMS Intervening Against Postoperative Delirium
Acronym: RECOVER
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: RenJi Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RECOVER
Record Dates: First submitted 2025-07-13; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Delirium
Keywords: cTBS; postoperative delirium; TMS; EEG
MeSH Terms: conditions — Emergence Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The effective coil or false coil shapes of the TMS group and the SHAM group were consistent. The assigned coils will blind clinical staff, patients, researchers, and outcome assessors who treat patients, and only data management personnel may unblind the assigned intervention measures. The statistical analysis of this experiment will be conducted using blinding, with the intervention group coded as (e.g. X and Y). Based on this blind analysis, two conclusions will be drawn: assuming X is the experimental group and Y is the control group, the other conclusion assumes the opposite. Two abstracts will be written and accepted by the author team. Afterwards, the blindness will be lifted.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TMS group (Experimental): The TMS group uses effective coils for transcranial magnetic stimulation treatment twice a day, with a treatment mode of continuous theta burst stimulation (cTBS). The stimulation intensity is set at 80% of the minimum exercise threshold.
  Interventions: Device: continuous Theta-burst stimulation
- SHAM group (Sham Comparator): For patients who experience postoperative delirium and are randomly assigned to the sham group, false coil stimulation is used. The auditory and scalp sensations induced by false coil stimulation are similar to those induced by effective coil stimulation, but there is no electromagnetic penetration into the brain or neural activation.
  Interventions: Device: Sham

INTERVENTIONS:
Device: continuous Theta-burst stimulation — Treatment parameters: each cTBS session consists of 50 Hz triplets of pulses delivered at 5 Hz for 40 s, totaling 600 pulses, and every set simulation includes 3 sessions. Electrodes are attached to designated head regions (right dorsolateral prefrontal cortex).
  Arms: TMS group
Device: Sham — the treatment mode was with sham coil.
  Arms: SHAM group

SUMMARY:
Postoperative delirium is common in elderly surgical patients and is associated with complications and prolonged hospitalisation. The aim of the RECOVER study is to assess the efficacy of electroencephalo graph (EEG)-transcranial magnetic stimulation (TMS) treatment for the management of postoperative delirium.

DETAILED DESCRIPTION:
Postoperative delirium(POD), a syndrome characterized by an acute change in attention, awareness and cognition, is one of the most common postoperative complications among elderly patients. Impaired neuronal network connectivity is likely one of the several neurobiological processes that contribute to POD pathogenesis. Recently, continuous theta burst stimulation (cTBS), a pattern of TMS, was demonstrated to improve cognitive function in patients with mild cognitive impairment.Recent research suggests that cTBS has positive effect on improving the connectivity and reorganization of the brain network.This project team conducted a pilot study in the early stage and innovatively applied cTBS to treat postoperative delirium in elderly patients. The results preliminarily elucidate the safety, and feasibility of TMS in treating postoperative delirium in elderly patients.

In order to confirm the effectiveness of EEG-TMS therapy for POD and observe its impact on long-term prognosis, this project will conduct a prospective randomized controlled study to compare TMS therapy with sham stimulation therapy. The study will observe The duration of postoperative delirium during the 7-day intervention period, as well as severity of delirium, the time to successful discharge (defined as the patient surviving outside the hospital for at least 48 hours after discharge), and the 30-day and 90-day survival times, the number of patients receiving salvage drug treatment, and the number of days each patient received salvage drug treatment, the sensitivity, specificity, and predictive value of EEG. The trial will provide new ideas for the prediction and treatment of postoperative delirium in clinic.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥60 years;
2. Scheduled for non-cardiac surgery;
3. Positive assessment for delirium via the CAM-ICU or 3D-CAM after surgery.

Exclusion Criteria:

1. Chronic use of antipsychotic medications;
2. Receipt of antipsychotic drugs prior to enrollment;
3. Permanently incapacitated patients (lacking decision-making capacity);
4. Inability to undergo delirium assessment (e.g., due to language barriers, deafness, blindness, aphasia, or coma);
5. Treatment withdrawal or brain death;
6. Known pregnancy or lactation;
7. Inability to obtain informed consent per national regulations;
8. Patients under compulsory hospitalization (involuntary commitment) by regulatory authorities;
9. Alcohol withdrawal delirium (delirium tremens);
10. Contraindications to transcranial magnetic stimulation (TMS);
11. Acute infectious diseases.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 98 (Estimated)
Dates: Start 2025-07-27 (Estimated); Primary Completion 2026-10-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Duration of postoperative delirium | 7 days
  Trained clinicians (who have received standardized CAM-ICU/3D-CAM training) will assess patients for POD using either the CAM-ICU or 3D-CAM tool twice a day.

SECONDARY OUTCOMES:
Severity of delirium | 7 days
  The severity of delirium is measured using the The Delirium Rating Scale-Revised-98 (DRS-R-98), which has a total score range of 0 to 46, with higher scores indicating greater severity of delirium.
Time to successful hospital discharge | 90 days
  Defined as discharge from the hospital with survival outside the hospital for ≥48 hours
Survival at 30 and 90 days | 90 days
  All-cause mortality
Number of patients receiving rescue medications | 7 days
  e.g., sedatives, antipsychotics, or other adjunctive therapies for delirium/agitation
Total days of rescue medication use per patient | 7 days
  Calculated as the sum of days each patient received such therapies

OTHER OUTCOMES:
Change from baseline on EEG | baseline, 7 days
  64-channel high-density EEG is used to assess the change of delta, theta, alpha, beta, gamma brainwave activity.
Change from baseline on sleep scales | Baseline, 90days
  The change is measured using the Pittsburgh Sleep Quality Index (PSQI), which provides a total score ranging from 0 to 21, with higher scores indicating worse sleep quality.
Change from baseline on stress scales | Baseline, 90days
  Stress is assessed using the Stress Appraisal Measure (SAM), which comprises six subscales rated on a 5-point Likert scale (1='not at all' to 5='extremely'). Higher scores on threat, centrality, and uncontrollability subscales indicate greater perceived stress, whereas higher scores on challenge, controllable-by-self, and controllable-by-others reflect lower stress.
Change from baseline on anxiety scales | Baseline, 90days
  Anxiety is assessed using the Generalized Anxiety Disorder-7 (GAD-7) scale, a 7-item self-report questionnaire where respondents rate symptom frequency over the past two weeks on a 4-point Likert scale (0="Not at all" to 3="Nearly every day"). The total score ranges from 0 to 21, with higher scores indicating greater anxiety severity.
Change from baseline on pain scales | Baseline, 90days
  The Short-form McGill Pain Questionnaire-2 (SF-MPQ-2) assesses pain intensity across 22 items (0-10 scale), with higher scores indicating worse pain.
Change from baseline on depression scales | Baseline, 90days
  The Patient Health Questionnaire-9 (PHQ-9) assesses depression severity through 9 items scored 0-3, with total scores ranging 0-27 (higher scores = worse symptoms).
Change from baseline on cognition scales | Baseline, 90days
  Cognition is assessed using the Montreal Cognitive Assessment (MoCA), a 30-point screening tool evaluating multiple domains (attention, memory, language, visuospatial skills), with higher scores indicating better cognitive function

CONTACTS AND LOCATIONS:
Locations (1):
- Renji hosipical, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided